CLINICAL TRIAL: NCT06580795
Title: How Can a Student Citizens' Assembly Facilitate the Co-creation of Nutrition Interventions in Higher Education Settings (DACCORD Study)
Brief Title: Co-creation of Nutrition Interventions in Higher Education Settings (DACCORD Study)
Acronym: DACCORD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Sorbonne Paris Nord (Other)
Collaborators: Paris 12 Val de Marne University (Other); National Research Agency, France (Other); Institute for Research in Public Health, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-055
Record Dates: First submitted 2024-08-23; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participation in the student citizens' assembly (Experimental): Participants are students participating in the student citizens' assembly
  Interventions: Behavioral: Student citizens' assembly

INTERVENTIONS:
Behavioral: Student citizens' assembly — The intervention consists in participating in a deliberative mini-public, a student citizens' assembly whose mission is to to co-create a list of concrete proposals that would improve the access of USPN students to sustainable diets and physical activity

SUMMARY:
The DACCORD study is a participatory research project which aims to provide insights on how to involve higher education students and diverse partners in the co-creation of campus nutrition interventions through a deliberative mini-public.

DETAILED DESCRIPTION:
The DACCORD study takes place at the University Sorbonne Paris Nord (USPN), located in the Seine Saint Denis department, in the Northern area of the Paris region (France). The intervention consists in a deliberative mini-public, a student citizen's assembly on diet and physical activity. The mandate of this student citizen's assembly is to co-create a list of concrete proposals that would improve the access of USPN students to sustainable diets and physical activity. The mini-public includes 30 students enrolled at USPN at the time of the study and a team of academic and non-academic partners involved in student life, nutrition, physical activity, or public policies.

The specific aims of the DACCORD study are 1) to design and implement a student citizens' assembly using participatory approaches, 2) to describe its process and evaluate its transferability, 3) to evaluate changes in nutritional habits, knowledge and citizen practices among students participating in the student citizen's assembly, using quantitative and qualitative methods.

Transferability will be evaluated continuously throughout the study, up to one year after completion of the student citizens' assembly. Nutritional habits, knowledge and citizen practices will be evaluated before and 1 months after the student citizens' assembly.

ELIGIBILITY:
Inclusion Criteria:

* being an adult (18 years of age or older)
* being enrolled at USPN at the time of the study
* being enrolled in initial training with in-person classes

Exclusion Criteria:

* being enrolled in continuing education or work-study programs

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Transferability indicators (Reach indicator of the RE-AIM framework) | Throughout implementation of the student citizens assembly (5 months)
  Proportion and representativeness of students participating in the mini-public
Transferability indicators (Effectiveness indicator of the RE-AIM framework) | Throughout implementation of the student citizens assembly (5 months)
  Qualitative analyses of the student citizens assembly proposals, in comparison with the recognized determinants of diet, using the DONE framework
Transferability indicators (Adoption indicator of the RE-AIM framework) | Throughout implementation of the student citizens assembly (5 months)
  Aggregated data on the characteristics of non-student members of the mini-public (in terms of gender, age, employer and job description)
Transferability indicators (Implementation indicator of the RE-AIM framework) | Throughout implementation of the student citizens assembly (5 months)
  Mini-public expertise, monetary cost of implementing the citizens' assembly, comparisont of actual vs. planned implementation
Transferability indicators (Maintenance indicator of the RE-AIM framework) | One year after completion of the student citizens assembly
  Qualitative evaluation of the actual implementation of the citizens assembly proposals and willingness of USPN representatives to replicate the student citizens' assembly in another location or on another topic (evaluated through individual interviews with USPN representatives)

SECONDARY OUTCOMES:
Changes in dietary habits | Before and one month after the student citizens' assembly
  Usual intake of the main food groups, assessed with a short food frequency questionnaire, and comparisons with current dietary recommendations
Changes in sustainable dietary practices | Before and one month after the student citizens' assembly
  Sustainable dietary practices (usual intake of plant-based and animal products, consumption of ultra-processed foods, usual intake of organic food, food supply locations, use of a composter, food waste and recycling, meal preparation habits), assessed with the SHED index. A higher score indicates greater sustainable practices.
Changes in knowledge of diet's environmental impact | Before and one month after the student citizens' assembly
  Knowledge of diet's environmental impact, assessed with a validated questionnaire. A higher score indicates greater knowledge.
Changes in citizens' practices | Before and one month after the student citizens' assembly
  Participation in civic activities (vote, forum, petition signing...), frequency of participation in online and offline political conversation, self-confidence when expressing opinions on diet, trust in the university institution, perceived usefulness of citizens' assemblies, assessed by questionnaire
Perception of the student citizens' assembly | Before and one month after the student citizens' assembly
  Motivations for participating in the student citizens' assembly, expectations on the role of this assembly, satisfaction with the proposals of the assembly, perceived quality of deliberations, assessed with an ad-hoc questionnaire
Academic-related data | Before the student citizens' assembly
  Study level (undergraduate, post-graduate, PhD student) and discipline
Changes in dietary habits and eating practices | Before the student citizens' assembly
  Changes in the interpretation of the term 'eating well,' understanding of the food system and its environmental impact, dietary habits and eating practices, barriers to sustainable diet, evaluated through semi-structured interviews
Socioeconomic status | Before the student citizens' assembly
  Scholarship status
Employment | Before the student citizens' assembly
  Employment status and weekly duration of job activities
Demographic characteristics | Before the student citizens' assembly
  Gender, accomodation type, commuting time between home and place of study, household cooking facilities

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bellicha, PhD, Principal Investigator — Université Sorbonne Paris Nord

IPD SHARING:
Plan to Share IPD: Undecided
Data described in the article, code book, and analytic code can be made available upon request. Researchers of a public institution can submit a collaboration request including their institution and a brief description of their project to the principal investigator. All requests will be reviewed by the steering committee of the Nutritional Epidemiology Research Team.

REFERENCES:
- [Derived] Bellicha A, Alles B, Baudry J, Boure L, Dehove H, El Karmouni H, Frenkiel E, Kesse-Guyot E, Peneau S, Mofakhami M; USPN Student Citizens' Assembly Group. A participatory research to assess how a student citizens' assembly can facilitate the co-creation of nutrition interventions in higher education settings. BMC Public Health. 2024 Oct 10;24(1):2772. doi: 10.1186/s12889-024-20277-3. PMID 39390476
- See also: Website of the student citizens' assembly — https://www.univ-spn.fr/convention-citoyenne-etudiante/